CLINICAL TRIAL: NCT01185730
Title: Evaluation of Prognostic Factors and Therapeutic Targets in Pulmonary Arterial Hypertension
Brief Title: Prospective Longitudinal Study of Patients With Idiopathic Pulmonary Arterial Hypertension, Family or Taking Anorectics
Acronym: EFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AOM 09065
Record Dates: First submitted 2010-08-05; First posted 2010-08-20 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Prognostic factors; Idiopathic pulmonary hypertension; Family pulmonary hypertension; use anorectics
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulmonary hypertension (Experimental): cohort of patients with pulmonary hypertension
  Interventions: Procedure: Right Heart Catheterization

INTERVENTIONS:
Procedure: Right Heart Catheterization — all patients of the all centers will have Right Heart Catheterization at the diagnosis

SUMMARY:
The objective of this clinical research is to analyze the survival of a cohort of patients newly diagnosed (incident cases) with idiopathic PAH, familial or associated with the use of anorectics (isolated pulmonary vascular disease without comorbidity) and identify prognostic factors using a dynamic model for predicting survival, including prognostic factors evaluated repeatedly at pre-specified periods during follow-up. In a second step, the investigators define using this model combinations of parameters to better define the therapeutic goals in PAH (functional class, exercise testing, hemodynamic, echocardiographic variables, biological parameters).

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare disease characterized by an intense proliferation of pulmonary arterial wall causing increased progressive pulmonary vascular resistance, leading to right heart failure and death. Established prognostic factors at diagnosis were identified 20 years ago at a time when there is no specific treatment for describing the natural history of disease.

Over the last 10 years, new therapeutic classes (similar to prostacyclin, antagonists of endothelin receptors, inhibitors of phosphodiesterase 5) have been developed and improved symptoms, exercise capacity, and hemodynamics in patients with PAH. With the availability of these new molecules, the clinician is now faced with difficult treatment decisions regarding the choice of initial treatment and the need for road treatments combined during evolution. Therapeutic purpose and effect of these different therapeutic strategies on the long-term survival remain poorly understood.

If it has been clearly demonstrated that clinical parameters (NYHA functional class), functional (test 6-minute walk) and hemodynamic (cardiac output and pulmonary vascular resistance) measured before initiation of treatment have a major role in determining the prognosis, with the contribution of new molecules is important to evaluate the prognostic value of changes in these factors during follow-up under specific treatment. At the baseline assessment, including repeat cardiac catheterization rights, it is also important to evaluate other prognostic criteria substitution, including methods of noninvasive evaluation (echocardiography, biomarkers).

ELIGIBILITY:
Inclusion criteria:

* Man or woman aged over 18 years
* With pulmonary arterial hypertension (PAH) idiopathic, hereditary or associated with the use of anorectics, newly diagnosed (less than 6 months) whose diagnosis was made by cardiac catheterization finding a mean pulmonary arterial pressure (mPAP)> 25 mm Hg at rest or> 30 mm Hg during exercise, with a pressure pulmonary artery occlusion (PAOP) ≤ 15 mm Hg,
* Has given his free and informed consent.

Exclusion criteria:

* Minor (age <18 years)
* PAH patients whose diagnosis was there more than 6 months (prevalent cases),
* Patient with PAH associated with concomitant disease (autoimmune disease, portal hypertension, HIV infection, congenital heart disease, schistosomiasis, chronic hemolytic anemia)
* Patient with veno-occlusive disease and / or pulmonary capillary hemangiomatosis suspected or documented
* Patients with pulmonary hypertension associated with left heart (pulmonary hypertension post-capillary)
* Patients with pulmonary hypertension associated with respiratory disease (chronic obstructive pulmonary disease, pulmonary fibrosis, sleep apnea syndrome Sleep)
* Patients with pulmonary hypertension post-embolic chronic
* Patient with pulmonary hypertension associated with sarcoidosis, histiocytosis X, a Lymphangioleiomyomatosis to mediastinal fibrosis,
* Adults protected
* Pregnant or lactating
* Persons deprived of liberty
* Persons in emergency situations,
* Persons who refused or unable to give informed consent.
* No affiliation to a social security scheme (beneficiary or beneficiary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
death frequency | 12 months

SECONDARY OUTCOMES:
death frequency | Evolution between baseline assessment and follow-up.
  A dynamic model for predicting survival will be used, including prognostic factors evaluated repeatedly at pre-specified periods during follow-up:
  * Right Heart Catheterization: mean pulmonary arterial pressure at rest or during exercise, and pressure pulmonary artery occlusion
  * Echocardiographic variables
  * Biomarkers (brain natriuretic peptide(BNP), N Terminal Pro BNP, Big-endothelin, Isoprostanes)
  * Functional Class of the New York Heart Association(NYHA)
  * Walk Test 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SITBON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France